CLINICAL TRIAL: NCT02389868
Title: Effects of Lovastatin on Human Platelet Proteome
Acronym: LovaC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Mathieu Fradet, MD/MSc student, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14221
Record Dates: First submitted 2015-03-05; First posted 2015-03-17 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Blood Platelets Proteome
Keywords: Lovastatin; Proteome; Blood platelets
MeSH Terms: interventions — Lovastatin

ARMS (1):
- Lovastatin (Experimental)
  Interventions: Drug: Lovastatin

INTERVENTIONS:
Drug: Lovastatin

SUMMARY:
The purpose of this study is to evaluate the effects induced by the cholesterol-reducing drug Lovastatin on the platelet proteome of healthy volunteers. Our results may allow to recognize the cell signalling modifications induced by Lovastatin. Furthermore, the current study aims to characterize the biological and inter-individual variation of platelet's proteome as measured by liquid chromatography-tandem mass spectrometry. Lastly, the exploration of changes induced by Lovastatin on the platelet's proteome may allow the discovery of modifications relative to the effects of statins on hemostasis and the lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* Being an individual age 18 to 40.
* If applicable, female participants susceptible of becoming pregnant consent to use a highly efficient contraception technique AND an efficient contraception technique during the clinical trial and at least 3 months following ending the consumption of Lovastatin.
* Being able to read and understand French.

Exclusion Criteria:

* Having a known history of dyslipidemia.
* In regard of the lipid profile at the first visit, patients that are not comprised between the 5th and the 95th percentile for LDL, HDL or Total cholesterol will be excluded.
* Having a history of hypersensitivity to Lovastatin, to one of the components of this product or to any other statin.
* Being affected by mental retardation.
* Pregnancy or suspicion of pregnancy.
* Having an excessive alcohol consumption (a maximum of 3 drinks a day during the trial will be accepted).
* Planning to perform unusual and very intense physical exercises during the study (ex: running a marathon or an Iron Man).
* Having a history of myopathy, myalgia or elevated creatine kinase (CK).
* In regard of the biochemical tests performed at the first visit, individuals having CK levels three times (or more) superior to the upper normal limit will be excluded.
* Having a personal or family history of hereditary muscular diseases.
* Having a history of renal or hepatic pathology.
* Taking one of the following drugs : any hypolipemic drug, any cytochrome P450 isoform 3A4 inhibitor (itraconazole, ketoconazole, posaconazole, voriconazole, HIV protease inhibitors, boceprevir, erythromycin, clarithromycin, telithromycin, nefazodone and products containing cobicistat), ACE inhibitors, danazol, verapamil, diltiazem, cyclosporin, amiodarone, colchicine, fusidic acid (IV or oral).
* Having a history of hypothyroidism.
* Having had a surgical intervention shortly before the beginning of the clinical trial.
* Suffering from any other acute medical condition.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Signal Intensity Measured for Each Protein Identified by Mass Spectrometry in Blood Platelets Lysates | Change from Baseline Protein Level at 6 Weeks
  Proteins from total platelets lysates will be analyzed by TripleTOF 5600 LC-MS/MS (AB SCIEX). The intensity measured for each identified protein will be recorded in SWATH mode. Intensities measured for each protein before (baseline) and after treatment with lovastatin (at 6 weeks) will be recorded and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche du CHUS, Sherbrooke, Quebec, Canada